CLINICAL TRIAL: NCT00876564
Title: Trauma System Evolution. A Quality Improvement Study of the Trauma System at Stavanger University Hospital, Norway.
Brief Title: Rogaland Trauma System Study
Acronym: RTSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Air Ambulance Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009/228-CAG(REK); 2009/228-CAG(REK)
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Trauma
Keywords: Triage precision
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trauma patients (Other): Included in trauma registry
  Interventions: Other: Trauma patients

INTERVENTIONS:
Other: Trauma patients

SUMMARY:
The purpose of this study is to improve performance, Stavanger University Hospital (SUH) reorganized key system structures and introduced in 2009 mandatory documentation of field Revised Trauma Score on trauma patients, tiered trauma team activation and new guidelines for field triage. Through a before and after study, the investigators aim to measure how the quality improvement initiative will influence structure, process and outcomes variables.

ELIGIBILITY:
Inclusion Criteria:

* Included in trauma registry

Exclusion Criteria:

* Excluded from trauma registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1812 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 7 years
  Over and undertriage

CONTACTS AND LOCATIONS:
Overall Officials: Marius Rehn, MD, Principal Investigator — Norwegian Air Ambulance Foundation
Locations (1):
- Stavanger University Hospital, Stavanger, Rogaland, Norway

REFERENCES:
- [Derived] Rehn M, Lossius HM, Tjosevik KE, Vetrhus M, Ostebo O, Eken T; Rogaland Trauma System Study Collaborating Group. Efficacy of a two-tiered trauma team activation protocol in a Norwegian trauma centre. Br J Surg. 2012 Feb;99(2):199-208. doi: 10.1002/bjs.7794. Epub 2011 Dec 20. PMID 22190166